CLINICAL TRIAL: NCT02553291
Title: A Clinical Trial of SystemCHANGE to Improve Exercise, Diet and Health in HIV-Infected Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Allison Webel, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CaseWestern
Record Dates: First submitted 2015-03-19; First posted 2015-09-17 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: HIV; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SystemCHANGE (Experimental): Subjects will participate in SystemCHANGE behavioral intervention focusing on diet and exercise. This six-session intervention focuses on system redesign of an individual's interpersonal environment and daily routines using small self-designed experiments to increase healthy behavior.
  Interventions: Behavioral: SystemCHANGE
- Control (Active Comparator): Subjects randomized to the control group will receive an usual care condition and pamphlets on diet and exercise from the U.S. Department of Agriculture and the American Heart Association (AHA)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: SystemCHANGE
  Other Names: BOBCAT Study
  Arms: SystemCHANGE
Behavioral: Control
  Arms: Control

SUMMARY:
HIV was once a fatal diagnosis, but due to treatment advances it is no longer a death sentence. Today, HIV-infected adults face a new challenge to their health; they are developing cardiovascular disease (CVD) earlier and more frequently than those not HIV-infected. Reasons for this include toxic effects of HIV medications and activation of the immune system. Preventing cardiovascular disease in HIV-infected adults will help them live healthier lives; however, there is a lack evidence to help us to achieve this goal. Exercise prevents cardiovascular disease, but it is often not addressed in HIV care, due, in part, to a lack of practical interventions targeting this population. This study will address this problem by testing an intervention to improve and maintain exercise in HIV-infected adults.

This study will examine the impact of an innovative and sustainable intervention, adapted to the unique medical and psychosocial needs of HIV-infected adults, called SystemCHANGE-HIV. It consists of six sessions to help redesign an individual's environment and routines to increase exercise.This is a randomized trial in which half of the subjects will participate in the intervention and half will participate in a control condition. Measures include assessments of exercise, fitness, and the markers of cardiovascular health before and after the intervention to see if, and how, they changed.

DETAILED DESCRIPTION:
Emerging evidence suggests that HIV infection is associated with a 1.5-2-fold higher risk of cardiovascular disease. This may be due, in part, to an increase in cardiometabolic risk factors related to the toxic effects of HIV medications, immune activation, and chronic inflammation. Interventions to prevent cardiovascular disease, accounting for the unique medical and psychosocial needs of HIV-infected adults, are needed.

Exercise has been shown to improve cardiometabolic risk and decrease cardiovascular disease. It has further been shown to improve cardiometabolic risk factors in some groups of HIV-infected adults in brief and intensely supervised trials. However, how to sustain exercise in this population with practical and scalable interventions that can be implemented in the home setting (i.e., free-living exercise) is unknown. The purpose of this is to test a novel, evidence-based intervention, SystemCHANGE-HIV, which holds promise for improving exercise in HIV-infected adults.

SystemCHANGE-HIV is a new behavior-change program that is based on a systems re-design model, in which the individual's daily routines are composed of a set of habits (behaviors) that can be changed. The intervention engages participants in a series of self-designed experiments to test ways to change their behaviors. The program involves six weekly group sessions to teach behavior-changing and exercise-improvement strategies, followed by monthly telephone booster sessions to encourage maintenance of beneficial effects. SystemCHANGE has significantly improved exercise adherence and cardiovascular risk factors in HIV-uninfected adults. The specific aims of our study are to (1) evaluate the 3-month and 6-month effects of SystemCHANGE-HIV on the amount and intensity of free-living exercise, and (2) describe the impact of SystemCHANGE-HIV on fitness (VO2 max) and cardiometabolic health.

To accomplish these aims, this is a longitudinal, randomized controlled trial (n=105) comparing the effects SystemCHANGE-HIV to those of an attention-control condition. The outcomes will be assessed for efficacy using biological and behavioral evaluations including: actigraphy, fitness assessments, and clinical laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

* aged >18 years
* have been diagnosed with HIV
* Receiving HIV antiretroviral therapy for at least 3 months
* have had at least one HIV viral load <400 copies/mL in the past 12 months
* at high lifetime risk for developing CVD (>females with >20% risk and males >30% risk using the Body-Mass Index (BMI) -based Framingham 30-year risk calculator)
* if on statin therapy, must have been on statins for the past 6 months

Exclusion Criteria:

* have an absolute or relative medical contraindication for exercise determined by the AHA criteria
* currently meet the Department of Health and Human Services recommendations for exercise (i.e.,150 minutes/week of moderate-intensity exercise or 75 minutes of vigorous-intensity exercise)
* have uncontrolled diabetes (HgA1c<8 at screening visit)
* are unable to understand spoken English
* expect to move out of the area within 12 months
* planning on becoming pregnant in the next six months
* are enrolled in a formal exercise, diet, or weight loss programs
* a household member who is or will be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Exercise as Measured by Waist-Worn Actigraph | 6 months
  Measured by Actigraph

SECONDARY OUTCOMES:
Cardiorespiratory fitness measured by VO2 max derived from a stress test | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Moore SM, Musil CM, Alder ML, Pignatiello G, Higgins P, Webel A, Wright KD. Building a Research Data Repository for Chronic Condition Self-Management Using Harmonized Data. Nurs Res. 2020 Jul/Aug;69(4):254-263. doi: 10.1097/NNR.0000000000000435. PMID 32205788
- [Derived] Moore SM, Musil CM, Jack AI, Alder ML, Fresco DM, Webel A, Wright KD, Sattar A, Higgins P. Characterization of Brain Signatures to Add Precision to Self-Management Health Information Interventions. Nurs Res. 2019 Mar/Apr;68(2):127-134. doi: 10.1097/NNR.0000000000000331. PMID 30540702